CLINICAL TRIAL: NCT01624584
Title: A Randomized-controlled Study Comparing Two Treatments for Children With Anxiety Disorders
Brief Title: A Study Comparing Two Treatments for Child With Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen Whiteside, PH D, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 11-008970
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety
Keywords: child; anxiety; CBT
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental treatment (Experimental): 6 sessions of anxiety treatment
  Interventions: Behavioral: Experimental treatment
- Traditional Treatment (Active Comparator): Six sessions of anxiety treatment
  Interventions: Behavioral: Traditional Treatment

INTERVENTIONS:
Behavioral: Experimental treatment — six sessions of child anxiety treatment
  Other Names: CBT; Cognitive behavioral therapy
  Arms: Experimental treatment
Behavioral: Traditional Treatment — six sessions of treatment consistent with current practice
  Other Names: CBT; Cognitive behavioral therapy
  Arms: Traditional Treatment

SUMMARY:
First, can exposure therapy for childhood anxiety begin earlier in the course of treatment than current treatment manuals suggest?

Second, is treating childhood anxiety with exposure therapy more effective and efficient than treating childhood anxiety with relaxation training + cognitive restructuring?

DETAILED DESCRIPTION:
Anxiety disorders are among the most common psychiatric disorders in children and typically produce significant disruption in family, social, and academic functioning (Merikangas & Avenevoli, 2002). Fortunately, treatments for childhood anxiety have been manualized and found to be efficacious (Walkup, et al., 2008). These treatments most often incorporate aspects of cognitive-restructuring, relaxation training, and exposure to anxiety-producing stimuli. Unfortunately, many practitioners opt to utilize mainly cognitive and relaxation techniques at the expense of exposure techniques (Freiheit, Vye, Swan, & Cady, 2004). However, it remains unclear which of these components is most effective in reducing anxiety symptoms or the extent to which they act in concert; thus, the relative effectiveness of treatment for childhood anxiety when leaving-out a treatment component is unknown. The current study aims to compare the relative effectiveness of exposure therapy for childhood anxiety to cognitive restructuring and relaxation techniques. Sixty children and adolescents seeking treatment for anxiety in an outpatient pediatric anxiety clinic will be randomized to receive either six sessions of parent assisted exposure therapy or six sessions of individual cognitive restructuring and relaxation training. Comprehensive assessments will be completed by trained clinicians at pre-treatment and again at post-treatment to measure reductions in anxiety and related symptoms as well as improvements in daily functioning. We anticipate that children treated with exposure therapy will demonstrate significantly greater improvement over the six sessions than children treated with cognitive-restructuring and relaxation training, and will require fewer additional treatment sessions. Support of this hypthothesis would clarify the active ingredients in manualized treatment for childhood anxiety disorders and would potentially lead to quicker, more efficient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have:

  1. a primary DSM-IV anxiety disorder diagnosis, including generalized anxiety disorder, obsessive compulsive disorder, panic disorder, separation anxiety disorder, social and specific phobias
  2. no medication changes were made at least 8 weeks prior to initiating participation in the study and during treatment.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  1. history of and/or current psychosis, autism, bipolar disorder, or current suicidality, oppositional defiant disorder, or eating disorder
  2. principal diagnosis other than one of the anxiety disorders listed for inclusion criteria
  3. current positive diagnosis in the child's caregiver of mental retardation, psychosis, or other psychiatric disorders or conditions that would limit his/her ability to understand CBT and follow-through with treatment directives.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale | Time 2
  Changes in PARS rating from time 1 to time 2 will be compared

SECONDARY OUTCOMES:
Pediatric Anxiety Rating Scales | Time 3
  Decrease in anxiety ratings from Time 1 to Time 3 will be compared between groups

OTHER OUTCOMES:
Attrition | Time 3
  Attrition in each condition will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Whiteside, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States